CLINICAL TRIAL: NCT00964106
Title: An Open-label Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Cytochrome P450 Probe Drugs in Healthy Adult Subjects
Brief Title: Validation Study of Multiple Probe Compounds for Drug Interaction Evaluation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 112684
Record Dates: First submitted 2009-07-23; First posted 2009-08-24 (Estimated); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Drug Interactions
Keywords: inducer; midazolam; inhibitor; rosiglitazone; dextromethorphan; caffeine; cocktail; pioglitazone; omeprazole; CYP; rosuvastatin; probe drug; drug interaction; flurbiprofen
MeSH Terms: interventions — Caffeine; Rosiglitazone; Flurbiprofen; Omeprazole; Dextromethorphan; Midazolam; Rosuvastatin Calcium; Ketoconazole; Fluconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probe drugs (Experimental): Caffeine 100 mg CYP1A2 Pioglitazone 15 mg CYP2C8 Flurbiprofen 40 mg CYP2C9 Omeprazole 20 mg CYP2C19 Dextromethorphan 45 mg CYP2D6 Midazolam 3 mg (Part 1, Part 2 Cohorts B and C)
  1 mg (Part 2 Cohort A) CYP3A4/5 Rosuvastatin 10 mg OATP1B1
  Interventions: Drug: Caffeine; Drug: Rosiglitazone; Drug: Flurbiprofen; Drug: Omeprazole; Drug: Dextromethorphan; Drug: Midazolam; Drug: Rosuvastatin
- Default Inhibitors (Experimental): A Ketoconazole 400 mg once-daily Day 1 through Day 9 CYP3A4 B Fluconazole 400 mg x1 dose on Day 1 200 mg once-daily Day 2 through Day 9 CYP2C9 C Rifampin 600 mg x1 dose on Day 1 and Day 8 OATP1B1
  Interventions: Drug: Ketoconazole; Drug: Fluconazole; Drug: Rifampin

INTERVENTIONS:
Drug: Caffeine — Caffeine dosed at 100 mg as probe for CYP1A2 pathway
  Arms: Probe drugs
Drug: Rosiglitazone — Dosed at 4 mg as probe for CYP2C8 pathway
  Arms: Probe drugs
Drug: Flurbiprofen — Dosed at 40 mg, probe for CYP2C9 pathway
  Arms: Probe drugs
Drug: Omeprazole — Dosed at 20 mg, probe for CYP2C19 pathway
  Arms: Probe drugs
Drug: Dextromethorphan — Dosed at 30 mg, probe for CYP2D6 pathway
  Arms: Probe drugs
Drug: Midazolam — Dosed at 3 mg for Part 1, Part 2 cohorts B and C and 1 mg for Part 2 Cohort A, probe drug for CYP3A4/5 pathway
  Arms: Probe drugs
Drug: Rosuvastatin — Dosed at 10 mg, probe drug for OATP1B1 pathway
  Arms: Probe drugs
Drug: Ketoconazole — Dosed at 400 mg once-daily Day 1 through Day 9, inhibitor of CYP3A4
  Arms: Default Inhibitors
Drug: Fluconazole — Dosed at 400 mg x 1 dose on day 1, 200 mg once daily on days 2 through 9, inhibitor of CYP2C9 pathway
  Arms: Default Inhibitors
Drug: Rifampin — Dosed at 600 mg x 1 dose on Day 1 and Day 8, inhibitor of OATP1B1 pathway
  Arms: Default Inhibitors
Drug: Rosiglitazone — Dosed at 15 mg, probe drug for CYP2C8 pathway
  Arms: Probe drugs

SUMMARY:
The purpose of this study is to identify and validate a probe cocktail for use in future drug-drug interaction studies. Cytochrome P450 enzymes and transport proteins play important roles in the disposition of drugs. Changes in the activity of these pathways can be assessed using probe drugs selected on the basis of their metabolic or transport pathway. This will be a two part study with the same subjects participating in both parts to decrease variability in data. The purpose of Part 1 is to identify a set of probe drugs ('cocktail') which do not interact with one another; groups of healthy volunteers will receive 7 probe drugs individually and as a combination of the 7 drugs given together as a cocktail. Part 2 will assess the performance of the probe cocktail using three known inhibitors (validation). The inhibitors plus probe cocktail will evaluate the ability of the newly established cocktail to accurately quantify metabolizing enzyme or transporter inhibition, representing a fundamental advance in probe cocktail validation and utility for drug development.

DETAILED DESCRIPTION:
The primary purpose of this study is to establish a validated drug cocktail, containing up to 7 probes, for assessing the activity of six drug metabolizing enzymes (CYP 1A2, 2C8, 2C9, 2C19, 2D6, 3A4/5) and the OATP1B1 transporter. In Part 1, the study will determine if there are pharmacokinetic interactions among the probe drugs by comparing the pharmacokinetics of the probe drugs when administered alone and in combination (i.e., as a cocktail). In Part 2, the study will evaluate the quantitative performance of the cocktail by examining the effect of select inhibitors on the pharmacokinetics of respective probe drugs when the probe drugs are administered alone versus when administered in the cocktail.

This study aims to establish a standard probe cocktail that can be used for drug-drug interaction studies, with the intention that any subset of the 7-drug cocktail could be selected for study with a drug in development.

In addition, this study will provide a proof-of-principle evaluation of dried blood spot technology as a method to measure drug concentrations in blood samples collected from clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician
* Subjects are not poor metabolizers based on genotyping for the major CYP2C9, 2C19, 2D6 alleles
* Male or female between 20 and 50 years of age at the time of screening, inclusive.
* A female subject is eligible to participate if she is of Non-childbearing potential or postmenopausal
* Body weight greater than or equal to 45 kg and BMI within the range 18.5 to 24.9 kg/m2 (inclusive).
* QTc < 450 msec
* Capable of giving written informed consent
* Able to understand and comply with protocol requirements

Exclusion Criteria:

* As a result of the medical interview, physical examination, or screening investigations, the Investigator considers the subject unfit for the study.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 7 days (14 days if the drug is a potential enzyme inducer, such as Panaz ginseng, Gingko biloba or St. John's Wort [Hypericum perforatum]) or 5 half-lives (whichever is longer) prior to the first dose of study medication. Herbal medications include, but are not limited to: traditional Chinese, Korean and Japanese medicines, Panaz ginseng, Gingko biloba or St John's wort (Hypericum perforatum) or any Traditional Chinese herbal medicines (TCM) South Asian Ayurvedic medicine, Traditional Korean Medicines and Japanese Kampo.
* Use of caffeine- or theobromine-containing beverages and foods, or alcohol-containing beverages within 72 hours prior to dosing
* Consumption of the following foods or drinks within 72 hrs prior to dosing : red wine, Seville oranges, grapefruits, pommelos, cruciferous vegetables (e.g., broccoli, Brussels sprouts, cabbage, celery), char-grilled meats, grapefruit juice.
* The subject has a positive pre-study drug/alcohol screen
* Urinary cotinine levels indicative of current smoking or history of regular use of tobacco- or nicotine-containing products within two months prior to screening.
* A positive Hepatitis B surface antigen or positive Hepatitis C antibody at screening.
* A positive test for HIV antibody
* History of regular alcohol consumption within 6 months of the study
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, five half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Systolic blood pressure outside the range of 80 to 140 mmHg, without antihypertensive therapy and no history of hypertension or diastolic blood pressure outside the range of 60 to 85 mmHg, or heart rate outside the range of 50 to 100 beats per minute (bpm) for female and 45 to 100 beats per minute (bpm) for male subjects
* History of syncope or vaso-vagal attacks.
* Pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic or renal function, that could interfere with the absorption, metabolism, or excretion of the study drugs.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Has a known intolerance or hypersensitivity to aspirin, NSAIDS, or benzodiazepines, or a known intolerance to the active and/or inactive ingredients in omeprazole, dextromethorphan, caffeine, rosiglitazone, pioglitazone, midazolam, rosuvastatin, flurbiprofen, ketoconazole, fluconazole, rifampin, quinidine, gemfibrozil, and fluvoxamine.
* Has any condition or symptom contraindicated for administration of the probe compounds or inhibitors
* History of sensitivity to heparin or heparin-induced thrombocytopenia (if heparin is used to maintain the patency of an intravenous cannula).
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* EGG abnormalities
* Pregnant females or lactating females.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2009-08-26 (Actual); Primary Completion 2011-08-29 (Actual); Study Completion 2011-08-29 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters | life of study
  Plasma AUC (0-inf) of probe and metabolite (where applicable) when administered alone, in combination with other probes/inhibitors

SECONDARY OUTCOMES:
To assess the safety and tolerability of co-administration of probe drugs | life of study
  Safety assessed by AE reporting, concurrent medication evaluation, clinical laboratory assessment, ECG, and vital sign assessment

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- South Korea (2):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 112684 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/112684?search=study&search_terms=112684#rs
- Available data/document: Study Protocol: 112684 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112684 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112684 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112684 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112684 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112684 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112684 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register